CLINICAL TRIAL: NCT01049464
Title: Efficacy of Magnesium Sulphate for Rate and Rhythm Control of New-onset Atrial Fibrillation in the Medical Critically Ill Patients: A Randomized, Controlled Trial
Brief Title: Magnesium Sulphate for Treatment of New Onset Atrial Fibrillation in Medical Intensive Care Unit Patient
Acronym: EMSAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Surat Tongyoo, Dr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si628/2009
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Hemodynamically unstable patients; Magnesium sulfate; Septic shock; Medical intensive care unit; New onset atrial fibrillation; Critically ill patients
MeSH Terms: conditions — Atrial Fibrillation; Shock, Septic | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5%D/W (Placebo Comparator): The patients in this group will receive 5%D/W 20 ml intravenous in 10 min and then 5%D/W 100 ml infusion in 6 hours as the placebo drug.
  Interventions: Drug: Placebo
- Magnesium sulphate (Experimental): The patients in this group will receive 2g of Magnesium sulphate diluted with 5%D/W into 20 ml solution, infusion intravenously in 10 min then 6g of Magnesium sulphate diluted with 5%D/W into 100 ml solution, infusion intravenously in 6 hours
  Interventions: Drug: Magnesium sulphate

INTERVENTIONS:
Drug: Placebo — 5%D/W 20 ml intravenous in 10 min then 5%D/W 100 ml intravenous in 6 hours.
  Other Names: 5%D/W
  Arms: 5%D/W
Drug: Magnesium sulphate — Magnesium sulphate 2g diluted with 5%D/W into 20 ml solution, intravenous infusion in 10 min then Magnesium sulphate 6g diluted with 5%D/W into 100 ml solution, intravenous infusion in 6 hours.
  Arms: Magnesium sulphate

SUMMARY:
The purpose of this study is to determine the efficacy of Magnesium sulphate for the rate and rhythm control of the new onset (within 48 hours) atrial fibrillation in the hemodynamically unstable patients, admitted in the medical intensive care unit patients.

DETAILED DESCRIPTION:
Atrial fibrillation is one of the most common arrhythmia, reported in the hemodynamically unstable patients in the intensive care unit. Loss of atrial contraction and the sequential atrioventricular contraction decrease the overall cardiac output which results in severe inadequate tissue perfusion. Medications aim for rate and rhythm control are recommended to treat new onset atrial fibrillation. These drugs (verapamil, diltiazem, amiodarone and beta blockers) may further compromise the patients' cardiac output by its' negative inotropic effect.

Magnesium sulphate with the cell membrane threshold potential stabilizing effect has been reported as an effective drug for rate and rhythm control for post-operative atrial fibrillation and the atrial fibrillation presented in the hospital emergency unit. However, there was inadequate data about the efficacy of Magnesium sulphate for treatment of new onset atrial fibrillation in the hemodynamically unstable patients admitted in the medical intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in medical intensive care unit
* Age 18 years or more
* New onset atrial fibrillation (within 48 hours), persist for at least 1 hour, ventricular rate 120 beats per min or more without evidence of volume depletion (CVP 8 mmHg or more or receive volume resuscitation about 20-30 ml/kg), oxygen saturation not less than 90%, serum Potassium level between 3.0-5.0 mEq/l, serum Calcium level between 8.0-11.0 mg/dl

Exclusion Criteria:

* Chronic atrial fibrillation
* Severe valvular heart disease including severe mitral regurgitation, mitral stenosis, aortic regurgitation, aortic stenosis, tricuspid regurgitation, tricuspid stenosis, pulmonic regurgitation or pulmonic stenosis
* Indicated for electrical cardioversion
* Severe hypomagnesemia (serum Magnesium < 1.2 mg/dl)
* Severe hypermagnesemia (serum Magnesium > 5.0 mg/dl)
* Renal insufficiency with creatinine > 3.0 mg/dl without renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion to sinus rhythm and/or ventricular rate less than 120 beats per min | 6 hours

SECONDARY OUTCOMES:
Blood pressure, superior vena cava or mixed venous oxygen saturation, cardiac index, inotropic and vasopressors dosage | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand